CLINICAL TRIAL: NCT03860415
Title: Probiotics as Intestinal Decolonization of ESBL-producing Enterobacteriaceae; a Randomized, Single Blinded, Placebo Controlled Clinical Trial
Brief Title: Can Probiotic Vivomixx Eradicate Colonization With ESBL?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-678678
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Antibiotic Resistant Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Vivomixx
  Interventions: Dietary Supplement: Vivomixx
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx — Two months of 2 sachets vivomixx each morning and 2 sachets each night. Each sachet of viviomixx contains 450 billion live bacteria.
  Arms: Probiotic
Dietary Supplement: Placebo — Two months of 2 sachets placebo each morning and 2 sachets each night. Each sachet of placebo contains 450 billion live bacteria.
  Arms: Placebo

SUMMARY:
Can probiotic Vivomixx eradicate Extended Spectrum BetaLactam (ESBL) colonization in adult patients?

DETAILED DESCRIPTION:
Infections due to extended spectrum cephalosporin-resistant Enterobacteriaceae (ESCRE) are a widely recognized public health threat. The prevalence of ESCRE is comparably low in Sweden but is steadily increasing; approximately 5 % of Swedish inhabitants are carrying ESCRE in the gut. ESCRE can lead to infections mainly from urine, abdomen and blood. These infections can be problematic to treat with current available antibiotics and represent a clinical challenge for clinicians around the world with considerable mortality and morbidity. Risk factors for acquiring an ESCRE is e.g. antibiotic treatment, trips to high prevalence countries, family member with ESCRE etc.

The duration of ESCRE carriage is not known. One Swedish study showed that ESCRE carriage can continue despite antibiotic treatment and that false negative cultures in between positive cultures are common. Since few new groups of antibiotics have been developed in the last decades, infections due to ESCRE may be increasingly difficult to treat. The possibility of ESCRE decolonization is therefore a desirable aim, in particular the more virulent enterobacteriaceae strains leading to recurrent clinical infection episodes.

Probiotics are microorganisms marketed as useful bacteria effective locally in the gut. In recent years many studies have focused on potential health benefits in a range of different gastrointestinal diseases e.g. ulcerous colitis, Crohn's disease, antibiotic associated diarrhoea where probiotics potentially have a therapeutic role4. Smaller studies have shown that probiotics possibly can bind and eliminate enteric pathogenic bacteria5-6. A small in vitro study showed that probiotics can be effective against antibiotic resistant bacteria. Larger clinical treatment studies are needed.

ESCRE constitutes a clinical problem and is largely seen in Escherichia coli and klebsiella spp. The investigator's theory is that the probiotic Vivomixx can reject ESCRE and thus decolonize the gut. Vivomixx contains eight different strains of probiotics; Bifidobacterium breve, B. longum, B. infantis, Lactobacillus acidophilus, L. plantarum, L. paracasei, L. bulgaricus, Streptococcus thermophilus and has the best documentation in clinical studies for enteric diseases of today.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (more than three months) ESBL colonization of the same strain as determined by
* species, phenotype and antibiogram.
* Patients must be able to swallow sachets.
* Must be able to speak and understand Swedish.
* Must have a permanent residence in Sweden.
* Must be able to sign informed consent in Swedish.

Exclusion Criteria:

* Immunosuppression (i.e. chemotheraphy, treatment with TNF-alpha-inhibitors).
* In patient care.
* immunodeficiency
* psychiatric disorder
* alcohol or substance abuse
* dementia
* Invasive catheters.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of participants that have changed from ESBL-postitive to ESBL-negative. | After 12 months, the number of participants that have changed from ESBL-postitive to ESBL-negative will be assessed.
  Each patient included provides three faecal samples after the intervention which will be selectively cultured for ESBL. Rate of patients that have three negative ESBL cultures will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Oskar Ljungquist, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ljungquist O, Kampmann C, Resman F, Riesbeck K, Tham J. Probiotics for intestinal decolonization of ESBL-producing Enterobacteriaceae: a randomized, placebo-controlled clinical trial. Clin Microbiol Infect. 2020 Apr;26(4):456-462. doi: 10.1016/j.cmi.2019.08.019. Epub 2019 Sep 5. PMID 31494254